CLINICAL TRIAL: NCT07283055
Title: A Swiss Interprofessional Network for Reviewing Inappropriate Medication in Primary Care: a Pilot Study
Brief Title: A Swiss Interprofessional Network for Reviewing Inappropriate Medication in Primary Care
Acronym: SINERGIC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bern (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: SINERGIC_01
Record Dates: First submitted 2025-12-02; First posted 2025-12-15 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Medication Review; Primary Care
Keywords: Clinical pharmacist; Medication review; Pharmaceutical service; Interprofessionality
MeSH Terms: interventions — Medication Review

STUDY DESIGN:
Intervention Model Description: Pilot trial; Before/after comparison
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient with medication review (Other)
  Interventions: Other: Medication review

INTERVENTIONS:
Other: Medication review — * Step 1 (optional): Patients taking at least 10 chronic medications and experiencing adherence or side effect issues may benefit from a specialised consultation with a pharmacist.
  * Step 2: The pharmacist identifies any medication-related issues for each patient and discusses them directly with the general practitioner in order to agree on the necessary adjustments.
  * Step 3: During a medical appointment, the doctor and patient will decide together whether to implement the proposed changes.
  * Step 4: The pharmacist will follow up after a few days and then again after 3 months.

SUMMARY:
The aim of the SINERGIC pilot study is to assess the feasibility in the Swiss context of implementing interprofessional medication reviews between GP and pharmacists, as part of a shared decision-making process with patients. The acceptability and potential effectiveness of such an intervention will also be assessed.

This assessment will enable the investigators to take into account the determining factors for setting up a large-scale study to support the sustainable financing of this service in the long term.

DETAILED DESCRIPTION:
The ageing population is leading to an increase in the prevalence of chronic conditions among older adults, often resulting in excessive polypharmacy. Polypharmacy, as well as the prescription of high-risk medications in this population, exposes them to more adverse effects, which can lead to falls and hospitalisation. This problem is of concern to healthcare professionals, whether they be general practitioners (GP), who have an overview of medical records, or dispensing pharmacists, who have an overview of medication. In Switzerland, these two professions still operate often in isolation from each other, but genuine collaboration is essential if we are to improve and manage polypharmacy among the elderly and limit the risks. Medication reviews are recognised as promising strategies for improving the quality of prescribing in patients with multiple medications.

This pilot trial does not randomly select participants and does not include a control group. It is a hybrid study that aims both to test the effectiveness of the intervention and to prepare for its implementation.

The study plans to include at least 250 patients from three groups of general practices in different settings. Participants will be aged 65 or older, take at least five chronic medications, and suffer from at least three chronic conditions. Individuals living in medical institutions will not be included.

Intervention:

* Step 1 (optional): Patients taking at least 10 chronic medications and experiencing adherence or side effect issues may benefit from a specialised consultation with a pharmacist.
* Step 2: The pharmacist identifies any medication-related issues for each patient and discusses them directly with the general practitioner in order to agree on the necessary adjustments.
* Step 3: During a medical appointment, the doctor and patient will decide together whether to implement the proposed changes.
* Step 4: The pharmacist will follow up after a few days and then again after 3 months.

Main objective: To assess whether this service is feasible in the context of the study.

Secondary objectives: Measure whether the intervention is well accepted (questionnaires and interviews) by the patients and healthcare professionals involved.

Exploratory objectives: Study the impact of the intervention on the quality of drug treatments, patients' quality of life and drug costs.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 65 years old;
* Regular use of at least 5 medications (chronic treatments, > 3 months);
* Patients with a minimum of 3 chronic diseases;
* Regular follow-up in a GP practice taking part in the project;
* Adequate understanding of French.
* Written informed consent

Exclusion Criteria:

* Residence in an institution (residential care facility, nursing home, etc.) ;
* Cognitive impairment preventing understanding or obtaining informed consent;
* Any other clinical situation deemed incompatible with participation, as decided by the GP in charge.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants recruited and percentage of participants retained | End of the study, expected to be on average after 4-6 months
  To assess the ability to recruit patients and retain patients for the duration of the follow-up and, if necessary, to explore the causes leading to their exit from the study; Measure: percentage
Number of GPs recruited and percentage of GPs retained | End of the study, expected to be on average after 18 months
  To assess the ability to recruit patients and retain patients for the duration of the follow-up and, if necessary, to explore the causes leading to their exit from the study; Measure: percentage

SECONDARY OUTCOMES:
Score of participants' acceptability of the intervention (Patients Reported Experience Measures) | End of the study, expected to be on average after 4-6 months
  Patients' acceptability of the service is assessed using a questionnaire adapted from the Short Assessment of Patient Satisfaction (SAPS). This is a short, 6 to 7-item scale used to assess patients' perceptions of the effectiveness of their treatments, and can help identify ways of improving a practice or intervention and responding to patients' concerns. Scale from 1 to 5, with higher values representing higher acceptance
Score of the healthcare professionals' acceptability of the intervention | End of the study, up to 18 months
  GPs' acceptability of the service is assessed using an online questionnaire inspired by the Collaboration and Satisfaction About Care Decisions (CSACD) questionnaire and the Assessment of Interprofessional Team Collaboration Scale (AITCS-II). A 6-items scale from 1 to 5, with higher values representing higher acceptance
  Additional semi-structured interviews based on a convenience sample will be conducted with health care professionals taking part to the main study by a trained student, in order to explore the conditions for implementing this new service in ambulatory care.
Qualitative evaluation of healthcare professionals' acceptability | End of the study, up to 18 months
  Semi-structured interviews based on a convenience sample will be conducted with health care professionals taking part to the main study by a trained student, in order to explore the conditions for implementing this new service in ambulatory care.
  Free text, qualitative analysis
Number and percentage of clinically relevant drug related problems resolved | 3 months after medical consultation
  The quality of medication therapy is assessed using a composite criterion based on five types of clinically relevant DRPs, taken from the recommendations of Beuscart et al. These DRPs will be documented using the validated PharmDisc tool adapted to our context. These DRPs reflect the appropriateness of prescribing. Their high frequency reflects poor prescribing quality. In order to standardise their identification, clinical pharmacists will be trained and using a protocol. PIMs will be identified according to the EU(7)-PIM list, which is a Europe-wide list.
Amount of drug cost savings | 3 months after medical consultation
  Savings in drug costs (in CHF) calculated for medications that were modified following the medication review and maintained three months later. The cost difference will be estimated using the change in drug daily dose multiplied by the public price per unit.
Cost of the service | During interprofessional meeting between GP and pharmacist
  Median cost of the intervention (in CHF) is calculated as the time invested by healthcare professionals (GPs, pharmacists) to conduct it multiplied by their average hourly wage.
Score on health-related quality of life (Patient-Reported Outcomes Measures or PROMs) | 3 months after medical consultation
  PROMs will be collected using a questionnaire adapted from the iSIMPATHY project, incorporating the EQ-5D-5L. The questionnaire assesses several dimensions: mobility, usual activities, pain/discomfort, anxiety/depression, as well as the patient's priorities in relation to their medication. A convenience sample will be drawn up with a minimum of 10 patients per group of GP practices.
  A five-items scale from 1 to 3, with higher values representing worst clinical outcomes

OTHER OUTCOMES:
Number of DRPs identified | Evaluation of pharmacists clinical skills, End of the study, up to 18 months
  Number of DRPs identified comparatively to those identified by the expert panel.
  Measure : percentage
Number and percentage of clinically relevant pharmaceutical interventions | Evaluation of pharmacists clinical skills, End of the study, up to 18 months
  Percentage of interventions clinically relevant evaluated by a panel of expert based on a standardised scale from 1 to 100, with higher values meaning best clinical relevance

CONTACTS AND LOCATIONS:
Overall Officials: Camille Lanfranchi, MSc, Study Chair — University of Bern (BIHAM); Juliane Fringeli, MSc, Study Chair — University of Bern (BIHAM)
Locations (1):
- Institute of Primary Health Care (BIHAM), Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mallet L, Spinewine A, Huang A. The challenge of managing drug interactions in elderly people. Lancet. 2007 Jul 14;370(9582):185-191. doi: 10.1016/S0140-6736(07)61092-7. PMID 17630042
- [Background] Liew TM, Lee CS, Goh SKL, Chang ZY. The prevalence and impact of potentially inappropriate prescribing among older persons in primary care settings: multilevel meta-analysis. Age Ageing. 2020 Jul 1;49(4):570-579. doi: 10.1093/ageing/afaa057. PMID 32365168
- [Background] Cole JA, Goncalves-Bradley DC, Alqahtani M, Barry HE, Cadogan C, Rankin A, Patterson SM, Kerse N, Cardwell CR, Ryan C, Hughes C. Interventions to improve the appropriate use of polypharmacy for older people. Cochrane Database Syst Rev. 2023 Oct 11;10(10):CD008165. doi: 10.1002/14651858.CD008165.pub5. PMID 37818791